CLINICAL TRIAL: NCT02901665
Title: Impact of Increased Parent Presence in the NICU on Parent & Infant Outcomes
Brief Title: Impact of Increased Parent Presence in the Neonatal Intensive Care Unit on Parent & Infant Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Susan M Horner, MS, APN/CNS, RNC-NIC, Clinical Nurse Specialist - Developmental Specialist, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-15866 Horner
Record Dates: First submitted 2014-10-09; First posted 2016-09-15 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Family Relationship; Stress; Breastfeeding; Bottle Feeding; Complications
MeSH Terms: conditions — Breast Feeding; Bottle Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-FCC Intervention (No Intervention): Pre-intervention group. No intervention will be administered.
- Post-FCC Intervention (Active Comparator): Following unit-wide implementation of FCC intervention consisting of communicating to families an expectation that they spend 4 hours per day in the NICU with their infants.
  Interventions: Other: FCC intervention

INTERVENTIONS:
Other: FCC intervention — Communication to all NICU families that they should be in the NICU a minimum of 4 hours/day.
  Arms: Post-FCC Intervention

SUMMARY:
The purpose of this pilot study is to compare parent and infant outcomes and unit outcomes pre and post a planned unit-wide intervention aimed at increasing parent presence in the Neonatal Intensive Care Unit (NICU). The FCC intervention will consist of communicating an expectation that all NICU parents be present at minimum 4 hours/day versus the current practice of telling families to "come as much as they can" that has resulted in inconsistent parent presence.

DETAILED DESCRIPTION:
Family centered care (FCC) is becoming the standard of care in the Neonatal Intensive Care Unit (NICU) and many benefits of FCC programs are reported in the literature. However, the integration of FCC practices remains inconsistent in NICUs and many families do not fully access available FCC supports. As a result NICU families continue to report feelings of powerlessness, stress, depression and lack of confidence in their ability to care for their infants at home. Studies of increased family presence in the NICU (8hours/day and 24/hours/day) have reported promising results for infants and families, but these studies report on programs implemented outside of the US. It is not known whether a program requiring fewer hours/day of parent presence, which may be a better fit with current US family demographics and policies, would demonstrate similar benefits. The purpose of this pilot study is to compare parent and infant outcomes and unit outcomes pre and post a planned unit-wide intervention aimed at increasing parent presence in the NICU. The FCC intervention will consist of communicating an expectation that all NICU parents be present at minimum 4 hours/day versus the current practice of telling families to "come as much as they can" that has resulted in inconsistent parent presence. Following informed consent, data will be collected on up to 45 NICU infants and families pre- and post- the intervention for a total sample of up to 90. Infant measures will include Salivary Cortisol levels, Infant weight gain, Length of Stay and Feeding route at discharge as well as rates of Family Visiting, Traditional Holding, Kangaroo Care (KC), and Breastfeeding. Parent measures will include Salivary Cortisol Levels and reported stress using the Parent Stress Scale: NICU. Unit-wide data will also be collected pre- and post- the intervention. Unit wide measures will include rates of Visitation, KC, Breastfeeding, Nosocomial Infections, IV infiltrates, Medication Errors and Incident (SERS) report rates.

ELIGIBILITY:
Inclusion Criteria:

* Less than 2 weeks of age
* Must be admitted to NICU

Exclusion Criteria:

* Previously discharged home
* <28 weeks gestation
* Anticipated hospital stay > 3 months

Ages: 1 Day to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Parent Salivary Cortisols | Throughout duration of NICU stay, an expected average of 4 weeks
  Salivary Cortisol levels obtained at admission, every 4 weeks and at discharge
Parent Stress Scale: NICU | Throughout duration of NICU stay, an expected average of 4 weeks
  Measured at admission and discharge using validated Parent Stress Scale: NICU
Infant Salivary Cortisol | Throughout duration of NICU stay, an expected average of 4 weeks
  Measured at admission, every 4 weeks and at discharge

SECONDARY OUTCOMES:
Family Visiting Rate | Throughout duration of NICU stay, an expected average of 4 weeks
  Rate of family visiting in hours per week
Parent Kangaroo Care Rate | Throughout duration of NICU stay, an expected average of 4 weeks
  Rate of Kangaroo Care (skin to skin holding of infant by a parent) per week
Breastfeeding Rate | Throughout duration of NICU stay, an expected average of 4 weeks
  Rate of mother providing breast milk for her infant

OTHER OUTCOMES:
Length of Stay in days | Throughout duration of NICU stay, an expected average of 4 weeks
  infant length of stay in days in the NICU from admission to discharge
Infant weight gain in grams/day | Throughout duration of NICU stay, an expected average of 4 weeks
  Average weight gain in grams/day throughout NICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Horner, MS, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (2):
- United States (2):
  - Neonatal Intensive Care Unit, Children's Memorial Hospital, Chicago, Illinois
  - Ann & Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cooper LG, Gooding JS, Gallagher J, Sternesky L, Ledsky R, Berns SD. Impact of a family-centered care initiative on NICU care, staff and families. J Perinatol. 2007 Dec;27 Suppl 2:S32-7. doi: 10.1038/sj.jp.7211840. PMID 18034178
- [Result] Gooding JS, Cooper LG, Blaine AI, Franck LS, Howse JL, Berns SD. Family support and family-centered care in the neonatal intensive care unit: origins, advances, impact. Semin Perinatol. 2011 Feb;35(1):20-8. doi: 10.1053/j.semperi.2010.10.004. PMID 21255703
- [Result] Reynolds LC, Duncan MM, Smith GC, Mathur A, Neil J, Inder T, Pineda RG. Parental presence and holding in the neonatal intensive care unit and associations with early neurobehavior. J Perinatol. 2013 Aug;33(8):636-41. doi: 10.1038/jp.2013.4. Epub 2013 Feb 14. PMID 23412640
- [Result] Franck LS, Cox S, Allen A, Winter I. Measuring neonatal intensive care unit-related parental stress. J Adv Nurs. 2005 Mar;49(6):608-15. doi: 10.1111/j.1365-2648.2004.03336.x. PMID 15737221